CLINICAL TRIAL: NCT04362501
Title: Efficacy of Dupilumab for Patients With Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP): a Randomized Double Blind Placebo Controlled Phase II Study
Brief Title: Efficacy of Dupilumab for Patients With Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00229130
Record Dates: First submitted 2020-04-21; First posted 2020-04-27 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Sinusitis
Keywords: sinusitis; chronic; treatment; non-polyposis
MeSH Terms: conditions — Sinusitis; Bronchiolitis Obliterans Syndrome | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: double blind randomized placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dupilumab treatment group (Experimental): dupilumab treatment group
  Interventions: Biological: dupilumab
- placebo group (Placebo Comparator): placebo group
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: dupilumab — 300mg dupixent SC every two weeks for six months
  Other Names: Dupixent
  Arms: dupilumab treatment group
Drug: placebo — placebo SC injection every two weeks for six months
  Arms: placebo group

SUMMARY:
The overarching objective of this study is to determine the clinical effectiveness of dupilumab for the treatment of CRS that includes several potential disease endotypes with the exclusion of the nasal polyp cluster that has previously been determined. The additional information gained from secondary and exploratory outcomes will help provide important insight for applied research studies and may also provide practical guidance to clinicians on how to select patients for treatment.

DETAILED DESCRIPTION:
Approximately 12% of adults in the United States, United Kingdom and other industrialized nations suffer from chronic sinus disease. Corticosteroids and antibiotic regimens are often used to treat the condition but the level of evidence to justify this approach is limited and at best offers only a transient solution. Furthermore, adverse side effects from the use of long-term oral steroids and concerns about skewing of the mucosal microbiota from overuse of antibiotics make these options problematic.

Currently, there are insufficient options for the approximately 30 million patients in the US suffering from chronic sinus disease. Recent phase 3 clinical trials found that dupilumab, an anti-IL4α receptor monoclonal antibody, reduces symptoms and polyp size in individuals with CRS with nasal polyps (CRSwNP). Similarly anti-IL5 antibodies have also been shown to have modest efficacy in this group of patients. However, for the approximately 65% of individuals with non-polyp related chronic sinus disease, these agents were not evaluated and there remains few viable options for therapy.

Chronic rhinosinusitis is defined as symptoms of nasal obstruction, facial pain or pressure, and mucopurulent drainage for at least 12 weeks along with evidence of mucosal disease by radiographic evidence or rhinoscopy. At least ten endotypes have been described although there is considerable overlap in terms of mucosal morphology, allergic status, the presence of polypoid tissue, and expression of biomarkers such as cytokines, specific IgE and other proteins. It may be incorrect to assume that the effectiveness of dupilumab demonstrated for those suffering with nasal polyps is exclusive to this CRS cluster alone.

One aspect to explain the differential effects of certain drugs and biologics on the treatment of CRS relates to host nasal and sinus microbial environment. The microbiome of CRS patients has been found to have reduced diversity, increased bacterial populations, and ultimately to have less stable bacterial networks. This imbalance of the microbiome may be a potential cause for sinus inflammation. Studies have demonstrated that Propionibacterium acnes for example, acts as an important stabilizing organism in the bacterial networks. Removal of this bacterial species e.g. from antibiotic use, may allow for more pathogenic organisms such as Staphylococcus or Streptococcus to flourish leading to increased inflammation.

An example of how Staphylococcus aureus may increase inflammation is through the production of superantigen that is thought to skew nasal inflammatory responses towards a Th2 dominated disease endotype. Other groups, have concluded that the host mucosal microbiota helps predict disease severity and might also predict susceptibility to certain therapies. Indeed, treatment with certain antibiotics has shown to modulate mucosal bacterial populations leading to clinical improvement and reduced polyp formation in some patients. It is not known whether host microbial and inflammatory milieu adequately predicts polyp formation or helps predict treatment success in the presence of dupilumab. The current study will include investigation of this important exploratory outcome.

The investigators have previously shown that modulation of both the innate and adaptive immune responses can impact dendritic cell and basophil responses in vitro and that these changes correlate with treatment success of patients with chronic allergic rhinosinusitis. The investigators also more recently discovered that IL-4 and IL-13 secreted by human basophils upregulates CD20 (mannose receptor), CD23 (FcεRII) and pSTAT6 expression on monocytes, while also promoting CCL17 (TARC) production by these cells. Other investigators have shown that the mannose receptor on monocytes negatively modulates TLR-4 innate immune signaling on dendritic cells that in turn affects T-cell polarization and response to allergens. The investigators might expect dupilumab to help attenuate this pathway resulting in a reduction of local sIgE production in the mucosa for example. It is already known that dupilumab reduces the expression of other inflammatory mediators such as CCL17 in asthma and atopic dermatitis. These aspects will be examined in the exploratory investigations using cell culture assays, flow cytometry and immunofluorescence pre and post treatment.

The overarching objective of this study is to determine the clinical effectiveness of dupilumab for the treatment of CRS that includes several potential disease endotypes with the exclusion of the nasal polyp cluster that has previously been determined. The additional information gained from secondary and exploratory outcomes will help provide important insight for applied research studies and may also provide practical guidance to clinicians on how to select patients for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 with history of chronic sinusitis without polyps
* SNOT-22 score of at least 30 at baseline
* Bilateral Lund-Mackay CT score 4 or more and/or MLK endoscopy score 4 or more
* Blood eosinophil count of at least 300/ul and/or SPT positive to at least 5/30 allergens, or eosinophil less than 300/ul and SPT negative (Th2 low group).
* Prior oral steroid or antibiotic use is acceptable but not required for entry
* Informed Consent
* Effective birth control (with <1% failure rate), post menopausal or documented abstinence
* Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
* All male subjects who are sexually active must agree to use an acceptable method of contraception (condom or vasectomy) from V1-V16

Exclusion Criteria:

* Immunosuppression other than oral steroids in the past 3 months
* History of nasal polyps within the past 3 years or noted at screening by CT or endoscopy
* Acute sinusitis at the time of entry
* Acute fungal sinusitis at the time of entry
* Uncontrolled asthma
* Cystic fibrosis
* Primary immune deficiency including CVID
* Other; serious concomitant illness or sinus disease that the investigator determines to disqualify
* A history of known immunodeficiency disorder including HIV
* History of hepatitis B or C
* Primary ciliary dyskinesia (PCD)
* Use of any biologic medication within the last 5 months or 5 half-lives whichever is longer
* Receipt of any investigational non-biologic within 5 half-lives prior to visit 0
* Receipt of immunoglobulin or blood products within 30 days prior to V1
* Scheduled sinus surgery
* Significant structural abnormalities or severe septal deviation
* Symptomatic or untreated life threatening cardiopulmonary disorders
* History of cancer not in remission at least 5 years prior to the date informed consent
* Subjects who are febrile (≥38°C; ≥100.4°F);
* Untreated helminth parasitic infection within 24 weeks prior to informed consent
* Pregnant or nursing
* Any other medical illness that precludes study involvement
* History of anaphylaxis to any biologic therapy or vaccine
* The following medications are excluded:

  * Any type of anti-interleukin therapy (e.g. Omalizumab, benralizumab, dupilumab mepolizumab, reslizumab, lebrikizumab etc.) within the last 5 months or 5 half-lives whichever is longer
  * Receipt of any investigational non-biologic within 30 days or 5 half-lives prior to visit 0, whichever is longer.
  * Immunosuppressive medications such as methotrexate, azathioprine, cyclosporine, tacrolimus
  * Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
  * Daily high dose aspirin greater than 81mg daily
  * Allergen Immunotherapy during build-up phase during the last three months
  * Other medications that could interfere with the action of dupilumab or suppress eosinophils

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
SNOT-22 | Every two weeks for six months
  Sino-Nasal Outcome Test (SNOT-22) survey score after six months treatment (range 0-110). Higher score means worse symptoms.

SECONDARY OUTCOMES:
Mini-RQLQ | Every two weeks for six months
  Mini-RQLQ (Rhinoconjunctivitis Quality of Life) validated survey (0-84). Higher score means worse symptoms.
UPSIT | Every two weeks for six months
  University of Pennsylvania Smell Identification Test (UPSIT) smell test (0-40). Higher score means better sense of smell.
Rescue medication | Every two weeks for six months
  Rescue medication use of corticosteroids. Specifically, prednisone mg use total over six month period.
CT Score | Once at screening and then at six month final visit
  Sinus CT Lund-Mackay (LM) score (0-24). Higher score means larger polyps.
Rhinoscopy Score | Once at screening and then at six month final visit
  Rhinoscopy modified Lund-Kennedy (MLK) score (0-12). Higher score means worse sinus disease.
Drop out rate rate | Continuous during entire length of study which is three years.
  Number of patients who leave the study. Individual participants will be considered to have dropped out if they leave the study for any reason during the six month treatment period. A total count will be collected over the entire study length estimated to be three years. This number will be divided by the total enrollment number to determine the rate of drop out.
Adverse event rate | Continuous during entire length of study which is three years.
  Significant Adverse Reactions (SAE). Individual participants will be monitored for serious adverse events during the six month treatment period. A total count will be collected over the entire study length estimated to be three years. This number will be divided by the total enrollment number to determine the rate of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jody Tversky, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No